CLINICAL TRIAL: NCT00856882
Title: The Effects of Soy Protein and/or Isoflavones on Glycemic Control, Insulin Sensitivity and Cardiovascular Risk Factors-a Six Months RCT Among Postmenopausal Women
Brief Title: The Effects of Soy Protein and Isoflavones on Glycemic Control, Insulin Sensitivity and Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Other Study IDs: CUHK4450/06M
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes; Cardiovascular Risk
MeSH Terms: conditions — Diabetes Mellitus | interventions — Soybean Proteins; Isoflavones; Milk Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- soy protein and isoflavones (Experimental)
  Interventions: Dietary Supplement: soy protein; Dietary Supplement: isoflavones
- milk protein and isoflavones (Experimental)
  Interventions: Dietary Supplement: isoflavones; Dietary Supplement: milk protein
- milk protein only (Placebo Comparator)
  Interventions: Dietary Supplement: milk protein

INTERVENTIONS:
Dietary Supplement: soy protein
  Arms: soy protein and isoflavones
Dietary Supplement: isoflavones
  Arms: milk protein and isoflavones; soy protein and isoflavones
Dietary Supplement: milk protein
  Arms: milk protein and isoflavones; milk protein only

SUMMARY:
The investigators propose to perform a double-blind, randomized placebo-controlled trial to examine the hypothesis that soy protein with isoflavones could improve glycemic control, insulin sensitivity and decrease cardiovascular risk factors in postmenopausal women with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese menopausal women aged 46-70 years with prediabetes or early untreated diabetes

Exclusion Criteria:

* Women with breast, ovary or other cancers in recent 5-year
* Severe renal or liver dysfunction
* Women with androgen excess
* Smokers
* Current use or recent (3-month)use of any drug or treatment for glycemic control, lipid improvement, weight reduction; Subjects with known soy or milk allergy.

Ages: 46 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2008-04 (Actual)

REFERENCES:
- [Derived] Liu ZM, Ho CS, Chen YM, Woo J. Can soy intake affect serum uric acid level? Pooled analysis from two 6-month randomized controlled trials among Chinese postmenopausal women with prediabetes or prehypertension. Eur J Nutr. 2015 Feb;54(1):51-8. doi: 10.1007/s00394-014-0684-1. PMID 24659208
- [Derived] Liu ZM, Ho SC, Chen YM, Ho YP. A mild favorable effect of soy protein with isoflavones on body composition--a 6-month double-blind randomized placebo-controlled trial among Chinese postmenopausal women. Int J Obes (Lond). 2010 Feb;34(2):309-18. doi: 10.1038/ijo.2009.236. Epub 2009 Nov 17. PMID 19918248